CLINICAL TRIAL: NCT01991210
Title: A Randomized, Open-Label, Multicenter, Phase II Trial Evaluating the Safety and Activity of DNIB0600A Compared to Pegylated Liposomal Doxorubicin Administered Intravenously to Patients With Platinum-Resistant Ovarian Cancer
Brief Title: A Study of DNIB0600A in Comparison With Pegylated Liposomal Doxorubicin (PLD) in Participants With Platinum-Resistant Ovarian Cancer (PROC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The primary objective of PFS did not meet pre-specified criteria.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO28609; 2012-005776-34 (EudraCT Number)
Record Dates: First submitted 2013-11-15; First posted 2013-11-25 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — lifastuzumab vedotin; 1-dodecylpyridoxal

ARMS (2):
- DNIB0600A (Experimental): DNIB0600A will be administered on Day 1 of each cycle (1 cycle = 21 days) until significant toxicity, disease progression, or withdrawal from the study (overall up to approximately 2.5 years).
  Interventions: Drug: DNIB0600A
- PLD (Active Comparator): PLD will be administered on Day 1 of each cycle (1 cycle = 28 days) until significant toxicity, disease progression, or withdrawal from the study (overall up to approximately 2.5 years).
  Interventions: Drug: PLD

INTERVENTIONS:
Drug: DNIB0600A — DNIB0600A will be administered at a dose of 2.4 mg/kg IV every 3 weeks.
  Other Names: RO5541081
  Arms: DNIB0600A
Drug: PLD — PLD will be administered at a dose of 40 mg/m^2 IV every 4 weeks.
  Arms: PLD

SUMMARY:
This randomized, multicenter, open-label study will evaluate the safety and efficacy of DNIB0600A (RO5541081) in comparison with PLD in participants with PROC, primary peritoneal cancer or fallopian tube cancer. Participants will be randomized to receive either DNIB0600A 2.4 milligrams per kilogram (mg/kg) intravenously (IV) every 3 weeks or PLD 40 milligrams per meter-squared (mg/m^2) IV every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically documented epithelial ovarian cancer, primary peritoneal cancer, or fallopian tube cancer
* Advanced epithelial ovarian, primary peritoneal, or fallopian tube cancer that has progressed or relapsed during or within 6 months after the most recent treatment with a platinum-containing chemotherapy regimen and for whom PLD is appropriate therapy
* No more than 1 prior cytotoxic chemotherapy regimens for the treatment of PROC and not more than 2 total regimens (defined as any therapy [approved or investigational] with intent to treat the ovarian cancer)
* Adequate hematologic, renal and liver function
* Willing and able to perform a patient-reported outcome (PRO) survey (including the possibility of using an electronic PRO device)
* For women of childbearing potential, agreement to use 1 highly effective form of contraception as defined by protocol through the course of study treatment and for 6 months after the last dose of study treatment

Exclusion Criteria:

* Primary platinum-refractory disease defined as disease progression during or within 2 months of a first-line, platinum-containing chemotherapy regimen
* Anti-tumor therapy, including chemotherapy, biologic, experimental, or hormonal therapy, within 4 weeks prior to Day 1
* Palliative radiation within 2 weeks prior to Day 1
* Prior anthracycline therapy, including prior treatment with PLD (for example, Doxil®, Caelyx®, or Lipodox®) in any setting (for example, in combination with carboplatin or as a single agent)
* Prior treatment with NaPi2b or SCL34A2 targeted therapy
* Major surgical procedure within 4 weeks prior to Day 1
* Current Grade greater than (>) 1 toxicity (except alopecia and anorexia) from prior therapy or Grade >1 neuropathy from any cause
* Left ventricular ejection fraction defined by multigated acquisition (MUGA)/echocardiogram below the institutional lower limit of normal
* Evidence of significant, uncontrolled, concomitant disease that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease or significant pulmonary disease
* Known active infection, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (within 4 weeks prior to Cycle 1, Day 1)
* Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis
* Presence of positive test results for hepatitis B or hepatitis C as detailed in the protocol
* Known history of HIV seropositive status
* Other malignancy within the last 5 years, except for adequately treated carcinoma in situ of the cervix, squamous carcinoma of the skin, adequately controlled limited basal cell skin cancer, or synchronous primary endometrial cancer or prior primary endometrial cancer
* Untreated or active central nervous system metastases (progressing or requiring anticonvulsants or corticosteroids for symptomatic control)
* Pregnancy or breastfeeding
* Known history of NaPi2b deficiency (for example, congenital alveolar microlithiasis or testicular microlithiasis)
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* Metabolic dysfunction, physical examination finding, or clinical laboratory find giving reasonable suspicion of a disease or condition that contraindicated use of an investigational drug or may render the participant at high risk from treatment complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2014-02-06 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2016-08-17 (Actual)

PRIMARY OUTCOMES:
Progression-free Survival According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | From baseline up to disease progression or death within 30 days of last study drug administration (overall up to approximately 2.5 years)

SECONDARY OUTCOMES:
Percentage of Participants With Objective Response According to RECIST v1.1 | From baseline up to 30 days of last study drug administration (overall up to approximately 2.5 years)
Duration of Objective Response | From occurrence of a documented objective response until relapse or death from any cause (overall up to approximately 2.5 years)
Overall Survival (OS) | From baseline up to death from any cause (overall up to approximately 2.5 years)
Percentage of Participants With Adverse Events (AEs) | From baseline up to 30 days of last study drug administration (overall up to approximately 2.5 years)
Area Under the Concentration-time Curve (AUC) of DNIB0600A | Pre-DNIB0600A infusion, 30 minutes post infusion (infusion length=90 minutes) on Day 1 of each Cycle (1cycle=21 days) (overall up to approximately 2.5 years); Day 8 of Cycle 1; Day 15 of Cycles 1-4
Maximum Concentration (Cmax) of DNIB0600A | Pre-DNIB0600A infusion, 30 minutes post infusion (infusion length=90 minutes) on Day 1 of each Cycle (1cycle=21 days) (overall up to approximately 2.5 years); Day 8 of Cycle 1; Day 15 of Cycles 1-4
Clearance (CL) of DNIB0600A | Pre-DNIB0600A infusion, 30 minutes post infusion (infusion length=90 minutes) on Day 1 of each Cycle (1cycle=21 days) (overall up to approximately 2.5 years); Day 8 of Cycle 1; Day 15 of Cycles 1-4
Elimination Half-life (t1/2) of DNIB0600A | Pre-DNIB0600A infusion, 30 minutes post infusion (infusion length=90 minutes) on Day 1 of each Cycle (1cycle=21 days) (overall up to approximately 2.5 years); Day 8 of Cycle 1; Day 15 of Cycles 1-4
Volume of Distribution at Steady State (Vss) of DNIB0600A | Pre-DNIB0600A infusion, 30 minutes post infusion (infusion length=90 minutes) on Day 1 of each Cycle (1cycle=21 days) (overall up to approximately 2.5 years); Day 8 of Cycle 1; Day 15 of Cycles 1-4
Percentage of Participants With Anti-therapeutic Antibodies (ATAs) Against DNIB0600A | Pre-DNIB0600A infusion on Day 1 of Cycles 1-4 (1cycle=21 days), at approximately 15-30 days after last infusion administration (overall up to approximately 2.5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (36):
- United States (14):
  - St. Joseph'S Hospital & Medical Center, Phoenix, Arizona
  - HonorHealth Research Institute - Pima Center, Scottsdale, Arizona
  - University of California Irvine Medical Center, Orange, California
  - Florida Cancer Specialists., St. Petersburg, Florida
  - Hematology & Oncology Associates, Covington, Louisiana
  - Johns Hopkins Uni; Oncology Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Inst., Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Oklahoma University Health Sciences Center, Oklahoma City, Oklahoma
  - Northwest Cancer Specialists, P.C., Tualatin, Oregon
  - Magee Womens Hospital, Pittsburgh, Pennsylvania
  - Women & Infants Hospital, Providence, Rhode Island
  - Sarah Cannon Cancer Center, Germantown, Tennessee
- Belgium (2):
  - UZ Leuven Gasthuisberg, Leuven
  - CHU Sart-Tilman, Liège
- Canada (3):
  - London Regional Cancer Centre, London, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Chum Hopital Notre Dame; Centre D'Oncologie, Montreal, Quebec
- France (4):
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer Rhône Alpes, Lyon
  - Hôpital Européen Georges Pompidou, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Institut Gustave Roussy, Villejuif
- Poland (3):
  - Bialostockie Centrum Onkologi, Bialystok
  - Wojewodzkie Centrum Onkologii, Gdansk
  - Wojskowy Instytut Medyczny Centralny Szpital Kliniczny MON, Warsaw
- Spain (5):
  - Hospital Universitario Vall d'Hebron; Servicio de Neumologia, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
- United Kingdom (5):
  - Sarah Cannon Research Institute, London
  - Christie Hospital, Manchester
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - The Royal Marsden Hospital, Sutton
  - Royal Marsden NHS Foundation Trust, Sutton, Surrey

REFERENCES:
- [Derived] Newhouse R, Nelissen E, El-Shakankery KH, Rogozinska E, Bain E, Veiga S, Morrison J. Pegylated liposomal doxorubicin for relapsed epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Jul 5;7(7):CD006910. doi: 10.1002/14651858.CD006910.pub3. PMID 37407274
- [Derived] Banerjee S, Oza AM, Birrer MJ, Hamilton EP, Hasan J, Leary A, Moore KN, Mackowiak-Matejczyk B, Pikiel J, Ray-Coquard I, Trask P, Lin K, Schuth E, Vaze A, Choi Y, Marsters JC, Maslyar DJ, Lemahieu V, Wang Y, Humke EW, Liu JF. Anti-NaPi2b antibody-drug conjugate lifastuzumab vedotin (DNIB0600A) compared with pegylated liposomal doxorubicin in patients with platinum-resistant ovarian cancer in a randomized, open-label, phase II study. Ann Oncol. 2018 Apr 1;29(4):917-923. doi: 10.1093/annonc/mdy023. PMID 29401246